CLINICAL TRIAL: NCT01161914
Title: A Multi-national Randomized Double Blinded Phase III Study to Evaluate the Safety and Efficacy of ISU302(Imiglucerase for Injection) or Cerezyme in Patient With Type I Gaucher Disease
Brief Title: The Safety and Efficacy Study of ISU302 in Patient With Type I Gaucher Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Lee, JaeHeung, ISU ABXIS CO., LTD
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ISU302-2008
Record Dates: First submitted 2010-07-11; First posted 2010-07-14 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2010-07

CONDITIONS: Gaucher Disease
Keywords: Type I Gaucher
MeSH Terms: conditions — Gaucher Disease | interventions — imiglucerase

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cerezyme® (Active Comparator): 60 U/kg infusion (every 2 weeks for 24 weeks)
  Interventions: Drug: Cerezyme®
- ISU302 (Experimental): 60 U/kg infusion (every 2 weeks for 24 weeks)
  Interventions: Drug: ISU302

INTERVENTIONS:
Drug: Cerezyme® — administered by IV infusion for a dose of 60 U/kg
  Arms: Cerezyme®
Drug: ISU302 — administered by IV infusion for a dose of 60 U/kg
  Arms: ISU302

SUMMARY:
The purpose of this study is to compare and evaluate the efficacy and safety of ISU302, an investigational product, and Cerezyme®, comparator, for Type 1 Gaucher Disease patients

ELIGIBILITY:
Inclusion Criteria:

* The subjects have a diagnosis of Type I Gaucher Disease
* Subjects between 2 years old and 75 years old
* Subjects documented with glucocerebrosidase deficiency
* Subjects with splenomegaly (as indicated by CT volumetric analysis as 5 times over than the standard size (0.2% of total body weight in kilograms))
* A hemoglobin concentration level:Male > 12 years of age <12.0 g/dL Female>12 years of age<11.0 g/dL Child > 2 years of age and <12 years of age <10.5 g/dL
* Platelet count of < 120,000 / ㎣
* Treatment-naive to enzyme replacement therapy (ERT) or treatment- experienced subjects who have not received ERT in the 12 months before screening and antibody test result is negative
* Treatment naive to substrate reduction therapy (SRT) or treatment- experienced subjects who have not received SRT in the 12 months before screening
* Subjects or their spouses who provide consent to use one of following contraception methods, or women in menopause. (In this case, menopause is defined as a period after 12 months from the last menstruation)
* Condoms, sponge, foams, jellies, diaphragm, or intrauterine device (Spouse or patient who had vasectomy or tubal ligation/ hysterectomy)
* Total abstinence from sexual intercourse: Female patient using oral contraceptives must use other contraception method (barrier method) also during the trial period and after the completion of trial as well as up to 90 days from the conclusion of trial.
* The subject or their legal representative has signed the informed consent.

Exclusion Criteria:

* Treatment with any investigational product in 90 days before study entry
* Partial or total splenectomy
* Subjects who have a serious concurrent disease like infection or who abuse addictive drug and substances.
* Pregnant and/or breast-feeding women
* Presence of Hepatitis B surface antigen or Hepatitis C or the patients show positive reaction to human immunodeficiency virus (HIV) type1
* Subjects with a history of allergic reaction to Imiglucerase
* Subjects with a history of severe pulmonary hypertension caused by Gaucher Disease
* Any subject whom the investigator or the sub investigator considers as inad equate for this trial

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
change in splenic volume compared to baseline | one year
  Primary endpoints to demonstrate non-inferiority of ISU302 against Cerezyme® for change in splenic volume compared to baseline.

SECONDARY OUTCOMES:
change in organ parameters and biochemical value compared to baseline | one year
  * Change in splenic volume compared to baseline for all subjects enrolled
  * Change in hemoglobin concentration
  * Change in platelet counts
  * Change in liver volume compared to baseline
  * Change in range variation of liver function test (ALT/AST)
  * Change in skeletal status improvement level
  * Change in bone mineral density
  * Change in biomarkers (acid phosphatase, angiotensin-converting enzyme (ACE) and chitotriosidase)
  * After the 1st administration, to evaluate pharmacokinetic profile by glucocerebrosidase activity assay